CLINICAL TRIAL: NCT05916027
Title: iTAPP Study - Identification and Treatment of Alcohol Problems in Primary Care
Brief Title: Identification and Treatment of Alcohol Problems in Primary Care
Acronym: iTAPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: iTAPP project
Record Dates: First submitted 2022-10-05; First posted 2023-06-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Abuse Alcoholism; General Practice; Screening and Brief Intervention
Keywords: Primary Care; Screening; Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Each participating clinic serves as its own control and as control for active clinics, in the stepped-wedge design. All clinics are inactive (no intervention) during the baseline period of three months.
- Active (Active Comparator): Active clinics are trained in the intervention object (the 15-method) prior to switching to the active group. Clinics are enrolled as active clinics (intervention) in four steps (4-5 clinics in each step). The intervention is implemented into the clinic, and the staff are free to use the intervention in everyday work.
  Interventions: Behavioral: The 15-Method

INTERVENTIONS:
Behavioral: The 15-Method — The 15-Method is a Screening and Brief Intervention method for identifying and treating alcohol problems in primary care. The method combines evidence-based approaches from specialized addiction treatment with screening and readily available treatment options in general practice to help identify and treat alcohol problems. The 15-method is based on Motivational Interviewing, Cognitive Behavioral Therapy and utilizes the Alcohol Use Disorder Identification Test (AUDIT) as a screening tool. The 15-Method contains three flexible steps: Identification of clinical problem related to alcohol; feedback and clinical work-up as needed; treatment. Treatment includes structured consultations (maximum of four) with patient home-work assignments, and can be combined with pharmacological treatment for alcohol problems.
  Arms: Active

SUMMARY:
The Identification and Treatment of Alcohol Problems in Primary Care (iTAPP) Study is a pragmatic cluster randomized controlled intervention trial evaluating the effectiveness of the 15-Method as an identification and treatment tool for alcohol-related problems in Danish general practice. The 15-Method combines evidence-based approaches from specialized addiction treatment with screening and readily available treatment options in general practice to help identify and treat alcohol problems in a primary care setting. The method has shown promising results as a treatment tool in Sweden. A feasibility study of the 15-Method in Denmark suggested that the method can be implemented in Danish general practice.

The trial is led by the Unit for Clinical Alcohol Research at The University of Southern Denmark in collaboration with The Research Unit of General Practice Odense at The University of Southern Denmark.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Affiliated with the participating general practices

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients exceeding the Danish national low-risk alcohol consumption limits | Four times during trial: Baseline (spring 2023), summer 2023, winter 2023/spring 2024, follow-up (summer 2024).
  Using Timeline Follow Back one-week data from patient surveys. The Danish national low-risk alcohol consumption limit is maximum 10 standard units (1 unit = 12 grams of ethanol) per week and maximum 4 standard units on a single day. Patients are coded 1 (drinking above limits) or 0 (not drinking above limits).
Number of heavy drinking days per week in patients | Four times during trial: Baseline (spring 2023), summer 2023, winter 2023/spring 2024, follow-up (summer 2024).
  The number of heavy drinking days (HDD) per week is derived from the Timeline Follow Back one-week (range 0-7 HDD/week) in patient surveys. A HDD is defined as >4 standard units (1 unit = 12 grams of ethanol) on the same day. Is a sum of the number of days patients drink >4 standard units.

SECONDARY OUTCOMES:
Likelihood of alcohol use being addressed during a consultation in general practice | Data is collected from enrollment in trial until the end of the trail (January 2023-August 2024).
  The likelihood of consultations in which the topic of alcohol has been addressed. Alcohol related consultations are continuously registered in the patient filing system throughout the trial period. An alcohol related consultation is defined as a consultation registered with the ICD-10 code z006 and ICPC-2 code A97.
Frequency of use of biomarkers as a screening tool for harmful alcohol use | Data is collected 1 year prior to trial start/enrollment (January 2022-December 2023) and from enrollment in trial until the end of the trial (January 2023-August 2024).
  The frequency of use in general practice. Biomarkers as a screening tool for harmful alcohol use comprise Gamma-Glutamyltransferase (GGT) and Alanine-Aminotransferase (ALAT). Data is obtained from Danish registers. The use of biomarkers as screening tool in the practices will be analyzed, comparing baseline levels to active (post-implementation) levels.
Prescription rate of pharmacological treatment for alcohol problems | Data is collected 1 year prior to trial start/enrollment (January 2022-December 2023) and from enrollment in trial until the end of the trial (January 2023-August 2024).
  The prescription rate in general practice. Pharmacological treatment for alcohol problems comprise Disulfiram, Naltrexone, Acamprosate, and Nalmefene. Data is obtained from Danish registers. The prescription rate in the practices will be analyzed, comparing baseline levels to active (post-implementation) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Anette S Nielsen, Professor, Study Director — Unit of Clinical Alcohol Research, University of Southern Denmark; Jens Søgaard, Professor, Principal Investigator — Research Unit of General Practice Odense, University of Southern Denmark
Locations (1):
- Unit for Clinical Alcohol Research, Clinical Institute, University of Southern Denmark, Odense C, Fynen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scholer PN, Volke KH, Andreasson S, Rasmussen S, Sondergaard J, Nielsen AS. The identification and treatment of alcohol problems in primary care (iTAPP) study: protocol for a stepped wedge cluster randomized control trial testing the 15-method in a primary care setting. Addict Sci Clin Pract. 2024 Jun 13;19(1):49. doi: 10.1186/s13722-024-00474-6. PMID 38872214